CLINICAL TRIAL: NCT03446131
Title: Improved Training Program for Fall Prevention of War Fighters With Lower Extremity Trauma
Brief Title: Improved Training Program for Fall Prevention of War Fighters
Acronym: RapidRehab
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kenton R. Kaufman, Ph.D., P.E. Director Motion Analysis Laboratory, Mayo Clinic
Other Study IDs: RRII; W81XWH-15-2-0071 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-12-11; First posted 2018-02-26 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Limb Injury
Keywords: transfemoral amputation; limb salvage; bilateral amputation; Department of Defense; orthosis; prosthesis; rehabilitation; military treatment facilities; military; injured lower extremity; prevent falls; trauma lower extremity; service members; retired service members; active service members; unilateral lower extremity trauma; limb amputation; limb preservation; preserved limb; trips; slips; transtibial amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will train War Fighters with lower extremity trauma to decrease fall risk.

DETAILED DESCRIPTION:
Eligible active duty service members, retired or veterans who participated in rehabilitation programs at Department of Defense Advanced Rehabilitation Centers (Walter Reed National Military Medical Center, Center for the Intrepid-San Antonio Military Medical Center and/or the Naval Medical Center San Diego) will be considered for enrollment in this study. This study will look at service members who have undergone transfemoral, transtibial or bilateral lower extremity amputation or limb salvage procedures. Participants will receive fall prevention training on an instrumented treadmill (6, training sessions). Participants will receive three performance assessments:-immediately following completion of the treadmill training and at three and six months following the completion of the training. Post training, twice per month subjects will receive an email containing a follow up fall questionnaire monitoring if they have fallen and the circumstances surrounding their fall. If they do not have access to email, or if a timely response is not received from the email questionnaire which was sent out, subjects will be contacted by phone.

ELIGIBILITY:
Inclusion Criteria:

* Eligible active duty and retired service members and veterans with lower limb trauma
* Transfemoral amputation, transtibial amputation, bilateral amputation and or limb salvage
* Participated in conventional rehab at one of the following rehab centers: Walter Reed National Medical Center, Center for the Intrepid Brooke Army Medical Center, Naval Medical Center San Diego
* Community ambulator
* Prosthesis / Orthosis use daily
* Exclusion Criteria:
* Dysvascular disease
* Excessive pain
* Neuromuscular problems preventing the performance of study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study plans to recruit both male and female military beneficiaries with a unilateral or bilateral transtibial or transfemoral amputation or salvaged and preserved limbs. The subjects will be present or past patients in the Naval Medical Center San Diego, C5 Rehabilitation Program, Center for the Intrepid Rehabilitation Program or Walter Reed National Military Medical Center Rehabilitation Program. Subjects will be contacted by the respective site study coordinator and asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Trunk Position | Change from baseline at 0, 3, and 6 months after completing training
  Trunk Position (referenced to vertical) at recovery step completion
Change in Trunk Velocity | Change from baseline at 0, 3, and 6 months after completing training
  Trunk Velocity at recovery step completion

SECONDARY OUTCOMES:
Falls | Change from baseline at 0, 3, and 6 months after completing training
  Falls per month reported in the Prosthesis Evaluation Questionnaire - Addendum
FSST | Change from baseline at 0, 3, and 6 months after completing training
  Four-Square Step Test

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Center for the Intrepid Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armed Forces Health Surveillance Center (AFHSC). Medical evacuations from Operation Iraqi Freedom/Operation New Dawn, active and reserve components, U.S. Armed Forces, 2003-2011. MSMR. 2012 Feb;19(2):18-21. PMID 22372753
- [Background] Doukas WC, Hayda RA, Frisch HM, Andersen RC, Mazurek MT, Ficke JR, Keeling JJ, Pasquina PF, Wain HJ, Carlini AR, MacKenzie EJ. The Military Extremity Trauma Amputation/Limb Salvage (METALS) study: outcomes of amputation versus limb salvage following major lower-extremity trauma. J Bone Joint Surg Am. 2013 Jan 16;95(2):138-45. doi: 10.2106/JBJS.K.00734. PMID 23324961
- [Background] Gooday HM, Hunter J. Preventing falls and stump injuries in lower limb amputees during inpatient rehabilitation: completion of the audit cycle. Clin Rehabil. 2004 Jun;18(4):379-90. doi: 10.1191/0269215504cr738oa. PMID 15180121
- [Background] Pauley T, Devlin M, Heslin K. Falls sustained during inpatient rehabilitation after lower limb amputation: prevalence and predictors. Am J Phys Med Rehabil. 2006 Jun;85(6):521-32; quiz, 533-5. doi: 10.1097/01.phm.0000219119.58965.8c. PMID 16715022
- [Background] Miller WC, Deathe AB, Speechley M, Koval J. The influence of falling, fear of falling, and balance confidence on prosthetic mobility and social activity among individuals with a lower extremity amputation. Arch Phys Med Rehabil. 2001 Sep;82(9):1238-44. doi: 10.1053/apmr.2001.25079. PMID 11552197
- [Background] Hausdorff JM, Rios DA, Edelberg HK. Gait variability and fall risk in community-living older adults: a 1-year prospective study. Arch Phys Med Rehabil. 2001 Aug;82(8):1050-6. doi: 10.1053/apmr.2001.24893. PMID 11494184
- [Background] Hornbrook MC, Stevens VJ, Wingfield DJ, Hollis JF, Greenlick MR, Ory MG. Preventing falls among community-dwelling older persons: results from a randomized trial. Gerontologist. 1994 Feb;34(1):16-23. doi: 10.1093/geront/34.1.16. PMID 8150304
- [Background] Dite W, Connor HJ, Curtis HC. Clinical identification of multiple fall risk early after unilateral transtibial amputation. Arch Phys Med Rehabil. 2007 Jan;88(1):109-14. doi: 10.1016/j.apmr.2006.10.015. PMID 17207685
- [Background] Franchignoni F, Orlandini D, Ferriero G, Moscato TA. Reliability, validity, and responsiveness of the locomotor capabilities index in adults with lower-limb amputation undergoing prosthetic training. Arch Phys Med Rehabil. 2004 May;85(5):743-8. doi: 10.1016/j.apmr.2003.06.010. PMID 15129398
- [Background] van Velzen JM, van Bennekom CA, Polomski W, Slootman JR, van der Woude LH, Houdijk H. Physical capacity and walking ability after lower limb amputation: a systematic review. Clin Rehabil. 2006 Nov;20(11):999-1016. doi: 10.1177/0269215506070700. PMID 17065543
- [Background] Miller WC, Speechley M, Deathe B. The prevalence and risk factors of falling and fear of falling among lower extremity amputees. Arch Phys Med Rehabil. 2001 Aug;82(8):1031-7. doi: 10.1053/apmr.2001.24295. PMID 11494181
- [Background] Krimmer H, Wiemer P, Kalb K. [Comparative outcome assessment of the wrist joint--mediocarpal partial arthrodesis and total arthrodesis]. Handchir Mikrochir Plast Chir. 2000 Nov;32(6):369-74. doi: 10.1055/s-2000-10915. German. PMID 11189889
- [Background] Macefield VG. Physiological characteristics of low-threshold mechanoreceptors in joints, muscle and skin in human subjects. Clin Exp Pharmacol Physiol. 2005 Jan-Feb;32(1-2):135-44. doi: 10.1111/j.1440-1681.2005.04143.x. PMID 15730450
- [Background] Lin YT, Berger RA, Berger EJ, Tomita K, Jew JY, Yang C, An KN. Nerve endings of the wrist joint: a preliminary report of the dorsal radiocarpal ligament. J Orthop Res. 2006 Jun;24(6):1225-30. doi: 10.1002/jor.20166. PMID 16705705
- [Background] Lewallen RP, Johnson EW Jr. Fractures in amputation stumps: review of treatment of 16 fractures. Mayo Clin Proc. 1981 Jan;56(1):22-6. PMID 7453246
- [Background] PALMER I. Pathophysiology of the medical ligament of the knee joint. Acta Chir Scand. 1958 Aug 30;115(4):312-8. No abstract available. PMID 13582512
- [Background] Bedigrew KM, Patzkowski JC, Wilken JM, Owens JG, Blanck RV, Stinner DJ, Kirk KL, Hsu JR; Skeletal Trauma Research Consortium (STReC). Can an integrated orthotic and rehabilitation program decrease pain and improve function after lower extremity trauma? Clin Orthop Relat Res. 2014 Oct;472(10):3017-25. doi: 10.1007/s11999-014-3609-7. PMID 24744130
- [Background] Patzkowski JC, Blanck RV, Owens JG, Wilken JM, Blair JA, Hsu JR. Can an ankle-foot orthosis change hearts and minds? J Surg Orthop Adv. 2011 Spring;20(1):8-18. PMID 21477527
- [Background] Patzkowski JC, Blanck RV, Owens JG, Wilken JM, Kirk KL, Wenke JC, Hsu JR; Skeletal Trauma Research Consortium. Comparative effect of orthosis design on functional performance. J Bone Joint Surg Am. 2012 Mar 21;94(6):507-15. doi: 10.2106/JBJS.K.00254. PMID 22437999
- [Background] Panwalkar N, Aruin AS. Role of ankle foot orthoses in the outcome of clinical tests of balance. Disabil Rehabil Assist Technol. 2013 Jul;8(4):314-20. doi: 10.3109/17483107.2012.721158. Epub 2012 Oct 19. PMID 23078248
- [Background] Guillebastre B, Rougier P. [Effects of rigid-ankle and ankle-foot orthoses in the control of asymetrical undisturbed upright stance]. Ann Readapt Med Phys. 2007 Mar;50(2):70-7. doi: 10.1016/j.annrmp.2006.09.002. Epub 2006 Oct 12. French. PMID 17070953
- [Background] Guillebastre B, Calmels P, Rougier P. Effects of rigid and dynamic ankle-foot orthoses on normal gait. Foot Ankle Int. 2009 Jan;30(1):51-6. doi: 10.3113/FAI.2009.0051. PMID 19176186
- [Background] Owens JG. Physical therapy of the patient with foot and ankle injuries sustained in combat. Foot Ankle Clin. 2010 Mar;15(1):175-86. doi: 10.1016/j.fcl.2009.10.005. PMID 20189123
- [Background] Owens JG, Blair JA, Patzkowski JC, Blanck RV, Hsu JR; Skeletal Trauma Research Consortium. Return to running and sports participation after limb salvage. J Trauma. 2011 Jul;71(1 Suppl):S120-4. doi: 10.1097/TA.0b013e3182219225. PMID 21795870
- [Background] Ramstrand N and Ramstrand S. (2010). The effect of ankle-foot orthoses on balance - Asystematic Review. Journal of Prosthetics and Orthotics; 22(4S): p4-p23.
- [Background] Hijmans JM, Geertzen JH, Dijkstra PU, Postema K. A systematic review of the effects of shoes and other ankle or foot appliances on balance in older people and people with peripheral nervous system disorders. Gait Posture. 2007 Feb;25(2):316-23. doi: 10.1016/j.gaitpost.2006.03.010. Epub 2006 May 9. PMID 16687248
- [Background] Shumway-Cook A, Woollacott MH. (1995). Motor learning and recovery of function. InMotor Control: Theory and Practical Application (pp. 23-443). Baltimore, MD:Williams & Wilkens.
- [Derived] Acasio JC, Tullos ML, Mahon CE, Khatri BR, Kaufman KR, Dearth CL, Hendershot BD. A single-subject comparison of functional outcomes between lower limb salvage vs. transtibial amputation through sequential participation in a fall-prevention program. Prosthet Orthot Int. 2022 Dec 1;46(6):614-618. doi: 10.1097/PXR.0000000000000156. Epub 2022 Jun 7. PMID 36515906
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials